CLINICAL TRIAL: NCT02092701
Title: Effects of a One Year Cholecalciferol Supplementation on Bone Health and Muscle Strength in Adults During Post-burn Period
Brief Title: Effects of Cholecalciferol Supplementation on Bone Health and Muscle Strength in Adults During Post-burn Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Rousseau, MD, University of Liege
Allocation: Randomized | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HDB1
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Vitamin D; Burn Injury
MeSH Terms: conditions — Burns | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- cholecalciferol (Experimental)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol

SUMMARY:
Vitamin D has pleiotropic effects. Burn patients are at risk of hypovitaminosis D and may experience post-injury osteopenia and sarcopenia. Investigators hypothesized that vitamin D supplementation during one year can improve bone and muscle health in post-burn period.

ELIGIBILITY:
Inclusion Criteria:

* occurrence of injury between 2005 and 2011
* burn surface area (BSA) greater than 10%

Exclusion Criteria:

* Pregnancy, renal or liver failure, hypo or hyperparathyroidism, prior vitamin D substitution, treatment using systemic corticosteroids or antiepileptic drugs, regular exposure to ultraviolet B radiation (solarium), unstable cardiovascular disease or acute muscle or skeletal injury prohibiting physical exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
calcidiol blood concentration | at the end of the protocol (after one year)

SECONDARY OUTCOMES:
bone health | at the end of the protocol (after one year)
  bone formation and resorption markers (blood concentrations) bone mineral density measurement using dual energy X-ray absorptiometry
muscle strength | at the end of the protocol (after one year)
  Measurements of knee muscles strength on an isokinetic dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Burn Centre, Liège, Belgium